CLINICAL TRIAL: NCT00932477
Title: Safety and Tolerability of Artificial Tears in Dry Eye Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: AG9965-001
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Results first posted 2011-12-13 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Glycerol; Polysorbates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Artificial Tear Formulation 1 (Experimental): Formulation 1: Carboxymethylcellulose Sodium, Glycerin and Polysorbate 80, based artificial tear
  Interventions: Drug: Formulation 1: Carboxymethylcellulose Sodium, Glycerin and Polysorbate 80, based artificial tear
- Artificial Tear Formulation 2 (Experimental): Formulation 2: Carboxymethylcellulose Sodium, Glycerin and Polysorbate 80, based artificial tear
  Interventions: Drug: Formulation 2: Carboxymethylcellulose Sodium, Glycerin and Polysorbate 80, based artificial tear
- Glycerin and Polysorbate 80 based artificial tear (Active Comparator): Glycerin and Polysorbate 80 based artificial tear
  Interventions: Drug: Glycerin and Polysorbate 80 based artificial tear

INTERVENTIONS:
Drug: Formulation 1: Carboxymethylcellulose Sodium, Glycerin and Polysorbate 80, based artificial tear — 1 to 2 drops into each eye three times per day
  Arms: Artificial Tear Formulation 1
Drug: Formulation 2: Carboxymethylcellulose Sodium, Glycerin and Polysorbate 80, based artificial tear — 1 to 2 drops into each eye three times per day
  Arms: Artificial Tear Formulation 2
Drug: Glycerin and Polysorbate 80 based artificial tear — 1 to 2 drops into each eye three times per day
  Other Names: Refresh Dry Eye Therapy®
  Arms: Glycerin and Polysorbate 80 based artificial tear

SUMMARY:
The safety and tolerability of two new artificial tears will be compared to a currently-available artificial tear in subjects with dry eye. Each subject will receive all three products in a randomly assigned order. The subject will use one product at a time for a duration of one week before switching to the next assigned product.

ELIGIBILITY:
Inclusion Criteria:

* Mild, moderate or severe symptoms of dry eye

Exclusion Criteria:

* Uncontrolled systemic disease
* Contact lens wear
* Participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a 3-treatment, 3-period, 6-sequence crossover study. Each subject received all 3 products in a randomly assigned order. The subject used 1 product at a time for a duration of 1 week before switching to the next assigned product (e.g., with treatments A, B, and C, the sequences were ABC, ACB, BAC, BCA, CAB, and CBA).
Groups:
- Sequence ABC: Started with Treatment A: Artificial Tear Formulation 1 followed by Treatment B: Artificial Tear Formulation 2 followed by Treatment C: Glycerin and Polysorbate 80 based artificial tear
- Sequence ACB: Started with Treatment A: Artificial Tear Formulation 1 followed by Treatment C: Glycerin and Polysorbate 80 based artificial tear followed by Treatment B: Artificial Tear Formulation 2
- Sequence BAC: Started with Treatment B: Artificial Tear Formulation 2 followed by Treatment A: Artificial Tear Formulation 1 followed by Treatment C: Glycerin and Polysorbate 80 based artificial tear
- Sequence BCA: Started with Treatment B: Artificial Tear Formulation 2 followed by Treatment C: Glycerin and Polysorbate 80 based artificial tear followed by Treatment A: Artificial Tear Formulation 1
- Sequence CAB: Started with Treatment C: Glycerin and Polysorbate 80 based artificial tear followed by Treatment A: Artificial Tear Formulation 1 followed by Treatment B: Artificial Tear Formulation 2
- Sequence CBA: Started with Treatment C: Glycerin and Polysorbate 80 based artificial tear followed by Treatment B: Artificial Tear Formulation 2 followed by Treatment A: Artificial Tear Formulation 1
Period: Treatment 1
Arm/Group | Sequence ABC | Sequence ACB | Sequence BAC | Sequence BCA | Sequence CAB | Sequence CBA
Started | 7 | 8 | 9 | 7 | 8 | 8
Completed | 7 | 8 | 9 | 7 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment 2
Arm/Group | Sequence ABC | Sequence ACB | Sequence BAC | Sequence BCA | Sequence CAB | Sequence CBA
Started | 7 | 8 | 9 | 7 | 8 | 8
Completed | 7 | 8 | 9 | 7 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment 3
Arm/Group | Sequence ABC | Sequence ACB | Sequence BAC | Sequence BCA | Sequence CAB | Sequence CBA
Started | 7 | 8 | 9 | 7 | 8 | 8
Completed | 7 | 8 | 9 | 7 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All Study Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 47
Age, Customized [Number; unit: participants]
  <40 years | 7
  >=40 years | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Tolerability Questionnaire Mean Scores at 1 Week
Description: Tolerability Questionnaire mean scores at 1 week. The Tolerability Questionnaire includes 8 tolerability questions on selected performance measures. All questions are scored based on continuous visual analog scale from 0-100. The first 4 questions presented measure increasing tolerability where 0=worst and 100=best. The second set of 4 questions presented measure decreasing tolerability where 0=best and 100=worst.
Time Frame: 1 Week
Population: Safety population, which consisted of all patients who started the study (randomized) and received treatment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Artificial Tear Formulation 1 | Artificial Tear Formulation 2 | Glycerin and Polysorbate 80 Based Artificial Tear
Number analyzed (Participants) | 47 | 47 | 47
Scores on a scale
  How comfortable is drop in the eye? | 70.1 (30.01) | 70.7 (26.63) | 57.3 (31.40)
  How soothing is drop in the eye? | 65.1 (31.67) | 65.9 (27.68) | 53.4 (32.63)
  How moistening/lubricating is drop in the eye? | 68.0 (27.79) | 65.9 (28.41) | 57.4 (31.51)
  How clear is vision with drop in the eye? | 66.0 (30.91) | 61.1 (30.78) | 53.0 (30.87)
  How much stickiness with drop in the eye? | 24.6 (29.44) | 19.5 (23.82) | 31.4 (29.03)
  How much blur with drop in the eye? | 33.2 (29.88) | 32.4 (30.52) | 48.9 (30.83)
  How much burning/stinging with drop in the eye? | 14.8 (22.48) | 14.3 (22.40) | 27.9 (30.62)
  How much discomfort with drop in the eye? | 19.3 (24.84) | 18.9 (26.27) | 27.1 (28.57)

2. Secondary Outcome: Number of Patients With at Least One Severity Grade Increase in Biomicroscopy Findings at 1 Week
Description: Number of patients with at least one severity grade increase in biomicroscopy findings at 1 week. Eyes are examined with a special microscope (biomicroscopy), and findings scored using a 5-point scale (0=none, +0.5=trace, +1=mild, +2=moderate, +3=severe). An increase in severity grade indicates worsening.
Time Frame: 1 Week
Population: Safety population, which consisted of all patients who started the study (randomized) and received treatment.
Measure: Number; unit: Number of Patients
Arm/Group | Artificial Tear Formulation 1 | Artificial Tear Formulation 2 | Glycerin and Polysorbate 80 Based Artificial Tear
Number analyzed (Participants) | 47 | 47 | 47
Number of Patients
  Pterygium (cornea) | 1 | 0 | 0
  Punctate keratitis (cornea) | 0 | 1 | 2
  Vital dye staining of cornea present | 0 | 1 | 0

3. Secondary Outcome: Best-Corrected Visual Acuity (BCVA) Status at 1 Week
Description: BCVA status at 1 week reported as the number of patients whose scores were either "Better", "No Change", or "Worse" than their scores at baseline. The status was tabulated as number of lines read correctly at 1 week minus the number of lines read correctly at baseline. "Better" equals increase of 2 lines or more in at least 1 eye; "No Change" equals change between -2 to +2 lines in either eye; "Worse" equals decrease of 2 lines or more in at least 1 eye. BCVA is measured using a special eye chart and is reported as the number of lines (5 letters per line) read correctly.
Time Frame: 1 Week
Population: Safety population, which consisted of all patients who started the study (randomized) and received treatment.
Measure: Number; unit: Number of Patients
Arm/Group | Artificial Tear Formulation 1 | Artificial Tear Formulation 2 | Glycerin and Polysorbate 80 Based Artificial Tear
Number analyzed (Participants) | 47 | 47 | 47
Number of Patients
  Better | 0 | 0 | 0
  No Change | 46 | 45 | 46
  Worse | 1 | 2 | 1

4. Secondary Outcome: The Number of Ophthalmic Adverse Events at 1 Week
Description: The number of ophthalmic adverse events (AE) at 1 week. An ophthalmic AE is any unfavorable and unintended sign, symptom, or disease related to the eye which occurs during the use of the study investigational product
Time Frame: 1 Week
Population: Safety population, which consisted of all patients who started the study (randomized) and received treatment.
Measure: Number; unit: Number of adverse events
Arm/Group | Artificial Tear Formulation 1 | Artificial Tear Formulation 2 | Glycerin and Polysorbate 80 Based Artificial Tear
Number analyzed (Participants) | 47 | 47 | 47
Number of adverse events
  Eye pruritis (itching) | 0 | 0 | 2
  Abnormal sensation in eye | 0 | 0 | 1
  Erythema (redness) of eyelid | 0 | 0 | 1
  Eyelid irritation | 0 | 0 | 1

ADVERSE EVENTS:
Groups:
- Artificial Tear Formulation 1: Formulation 1 Carboxymethylcellulose Sodium, Glycerin and Polysorbate 80 based artificial tear
- Artificial Tear Formulation 2: Formulation 2 Carboxymethylcellulose Sodium, Glycerin and Polysorbate 80 based artificial tear
Arm/Group | Artificial Tear Formulation 1 | Artificial Tear Formulation 2 | Glycerin and Polysorbate 80 Based Artificial Tear
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo